CLINICAL TRIAL: NCT05039996
Title: Effectiveness of Integrated Education and Relaxation Program on Migraine Related Disability in Patients Attending Headache Clinic, Ain Shams University Hospitals: A Randomized Controlled Trial
Brief Title: Effectiveness of Education and Relaxation Program on Migraine Related Disability in Patients Attending Headache Clinic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMASU M D 231/2018
Record Dates: First submitted 2021-08-10; First posted 2021-09-10 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-08

CONDITIONS: Migraine Headache
Keywords: Migraine; Health Education; Relaxation Training; Disability
MeSH Terms: conditions — Migraine Disorders; Health Education | interventions — Educational Status; Relaxation Therapy

STUDY DESIGN:
Intervention Model Description: The participants in the intervention group will receive the education and training program in addition to the routine pharmacological treatment whereas the participants in the control group will receive only the routine pharmacological treatment.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Educational and training part. The educational part will be done once in the first visit in about 30 minutes Information and skills will be demonstrated and applied in the session through power point presentation, educational brochures, and video lessons and guided home-based practice.
  Appropriate relaxation training Program
  * Relaxation training comprises deep breathing exercises and progressive muscle relaxation, to perform them daily and to keep a record of them.
  * Group meeting sessions for training will be held every week for the 1st 4 weeks
  * Video programs will be used as relaxation facilitators.
  * Patient will try these exercises for the first time in front of the researcher.
  * Patients will be advised to perform them daily for 8 weeks to achieve 60 sessions and to keep a record of them.
  Follow up of the intervention group adherence to instructions will be done weekly by Telephone.
  Interventions: Behavioral: education and relaxation program
- Control group (Placebo Comparator): The control group will be advised to be adherent to the prescribed medications only and try not to change the treatment plan during the study period.
  Interventions: Behavioral: education and relaxation program

INTERVENTIONS:
Behavioral: education and relaxation program — randomized controlled trial
  Other Names: integrated therapeutic patient education and relaxation program

SUMMARY:
Migraine causes severe impairment in quality of life (QOL) both during and between attacks. Migraine also increases absenteeism, reduces productivity at work as well as at home, disrupts social and family relationships, also is associated with increased healthcare costs.

The current study aiming to evaluate the effectiveness of an integrated therapeutic patient education and relaxation training intervention in order to decrease the burden of migraine headache among adult patients attending the headache clinic in Ain Shams University Hospitals.

DETAILED DESCRIPTION:
- The participants will be assessed for their eligibility based on inclusion and exclusion criteria. After obtaining the written informed consent, the eligible participants will be randomized to either an intervention or a control group. Psychiatric and personality disorders will be excluded before participation using the translated form of (Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders) I and II questionnaires.

The participants in the intervention group will receive the education and training program in addition to the routine pharmacological treatment whereas the participants in the control group will receive only the routine pharmacological treatment (preventive treatment with stable dose for at least 3 months and not to change the dose through the study).

For proper conduction of the study, three phases will be performed:

Assessment phase:

Each migraine patient in the intervention and control group will be interviewed individually before applying the planned program to collect socio-demographic data and clinical migraine evaluation using the clinical sheet of the clinic. Then base line measures of headache-related disability and migraine specific quality of life using migraine specific quality of life questionnaire before any intervention. Retrospective recording of 1 month past migraine attacks frequency will be recorded. This interview will take about 25-30 minutes.

Implementation phase:

* intervention group An intervention program will be implemented to the intervention group only after dividing them into small homogeneous groups. The program will be conducted in the clinic, it includes two parts educational and training part.

The educational part will be done once in the first visit in about 30 minutes aiming to increase patient knowledge about migraine reduce the impact of migraine in daily life, the session will include concise messages about:

1. Basic migraine education.
2. Identify Common triggers to reduce and avoid migraine attacks.
3. Role of non-pharmaceutical therapies.
4. Steps for getting support from family, friends and at work.
5. Encourage use of the headache dairy.
6. How to prepare migraine emergency tool kit.
7. Explanation and demonstration of progressive muscle relaxation and deep breathing training (20-30min).

Information and skills will be demonstrated and applied in the session through power point presentation, educational brochures, video lessons and guided home-based practice.

The information will be in a simple language, relevant to the disease process and management as well as evidence-based (guidelines for controlled trial in migraine, 2012).

The practical part:

Appropriate relaxation training Program

* Relaxation training comprises deep breathing exercises and progressive muscle relaxation, to perform them daily and to keep a record of them.
* Group meeting sessions for training will be held every week for the 1st 4 weeks .
* Video programs will be used as relaxation facilitators.
* Patient will try these exercises for the first time in front of the researcher.
* Patients will be advised to perform them daily for 8 weeks to achieve 60 sessions and to keep a record of them.

Follow up of the intervention group adherence to instructions will regularly be done weekly by Telephone for the remainder of the study between educational, reinforcement and final evaluation sessions.

Participants who will return for reinforcement sessions will receive mild compensation for study participation.

The control group The control group will be advised to be adherent to the prescribed medications only and try not to change the treatment plan during the study period.

Evaluation phase:

Evaluation of both groups will be done using headache diary and migraine specific quality of life questionnaires. After another 4 weeks, the two groups' participants will be reevaluated. Final evaluation will be done after 3 month from base line by the researcher using the same tools.

•Statistical Analysis /Statistical Package:-

-The data will be collected, revised, coded and entered to personal computer, Statistical analysis by the appropriate statistical tests will be done using (statistical package for social science) program version 20.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years old.
* Diagnosed with migraine for at least 6 months duration.
* Experiencing 4 or more migraine days/month with disability.
* Willingness to practice relaxation exercises at home.

Exclusion Criteria:

* Secondary headache.
* Patients with severe co-morbid psychiatric (depression, anxiety), personality or medical condition (liver or renal impairments).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the intervention program on headache frequency | 3 month
  Attacks frequency, expressed in days per month , will be collected from the "headache diary" filled in by the patient.
  Data will be recruited from the diary at base line and after another 4 weeks, Final evaluation will be done after 3 month
Effectiveness of the intervention program on headache intensity | 3 month
  The average of monthly attacks intensity ( severity) will be measured using the (Numerical rating scale) (from 0 to 10 scales) included in the headache diary Data will be recruited from the diary at base line and after 4 weeks, Final evaluation will be done after 3 month from beginning of the intervention program
Effectiveness of the intervention program on headache (attacks) duration | 3 month
  The average of monthly attacks duration will be calculated from the headache diary filled in by the patient at base line,4 weeks and finally after 3 month from the baseline evaluation

SECONDARY OUTCOMES:
Effectiveness of the intervention program on headache related quality of life and disability | 3 month
  By using the "Migraine specific quality of life questionnaire (MSQ)": The MSQ is a 14-items measure designed to assess the effects of migraine on an individual's quality of life. There are three MSQ subscales, Emotional (MSQ-E), restrictive (MSQ-R), and preventive (MSQ-P). The MSQ is a reliable and valid questionnaire in migraine patients that can determine the functional impact of migraine.
  Evaluation of both groups will be done using "MSQ questionnaire" at base line and after another 4 weeks, Final evaluation will be done after 3 month from base line by the researcher using the same tool.

CONTACTS AND LOCATIONS:
Overall Officials: Sara H Abd El Khalek, Principal Investigator — Assistant lecturer ,Family medicine department; Ayat F Mohamed, Study Chair — lecturer,Community, Environmental and Occupational medicine; Randa M Amin, Study Chair — lecturer in neurology department; Mohammed M Fouad, Study Chair — Assistant professor, neurology department; Diaa M Abd El Hamid, Study Chair — Head of Family Medicine Department.; Hisham A Hatata, Study Chair — professor psychiatry department
Locations (1):
- Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
individual participant data that underlie the results reported in this article
Supporting Information: Study Protocol, SAP
Time Frame: beginning 3 month and ending 7 years following article publication
Access Criteria: proposals should be directed to the chief author

REFERENCES:
- [Background] Tfelt-Hansen P, Pascual J, Ramadan N, Dahlof C, D'Amico D, Diener HC, Hansen JM, Lanteri-Minet M, Loder E, McCrory D, Plancade S, Schwedt T; International Headache Society Clinical Trials Subcommittee. Guidelines for controlled trials of drugs in migraine: third edition. A guide for investigators. Cephalalgia. 2012 Jan;32(1):6-38. doi: 10.1177/0333102411417901. No abstract available. PMID 22384463
- [Background] Eghbal Sekhavati, Mojtaba Rahimian Boogar, Rouhi Afkari, Somayeh Kasharafifard, Vahideh Parsaei Mehr, Fatemeh Lotfi Mola and Kobra Ahanijegar, 2016. The Study of the Effectiveness of Progressive Muscle Relaxation to Reduce Symptoms in Women with Migraine Headache. Research Journal of Medical Sciences, 10: 175-184.